CLINICAL TRIAL: NCT03837496
Title: Symptom-Targeted Randomized Intervention for Distress and Adherence to Adjuvant Endocrine Therapy (STRIDE) Among Breast Cancer Survivors: A Pilot Feasibility Trial
Brief Title: Small-group, Virtual Program for Improving Symptoms and Distress Related to Hormonal Therapy for Breast Cancer Survivors
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jamie Jacobs, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-603; K07CA211107 (NIH)
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Adherence, Medication
Keywords: Breast Cancer; Endocrine Therapy; Hormonal Therapy; Symptoms; Distress; Survivors
MeSH Terms: conditions — Breast Neoplasms; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the participant's study condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STRIDE Run-In (Experimental): * Stride is delivered as a Five weekly one-hour virtual (videophone) or in-person sessions in small groups with a trained clinician
  * Two 15-minute check-in phone calls later in the study
  * Participants will store hormonal therapy medication in a bottle provided by the study team.
  * Participants will complete questionnaires at enrollment and 3-months post- enrollment
  Interventions: Other: STRIDE
- STRIDE (Experimental): * Stride is delivered as six weekly one-hour virtual (videophone) sessions in small groups with a trained clinician (or individually, in the rare instance in which scheduling doesn't allow for groups and the participant is approaching the 12-week assessment window)
  * Two 15-minute check-in phone calls later in the study
  * Participants will store hormonal therapy medication in a bottle provided by the study team.
  * Participants will complete questionnaires at enrollment, 12-weeks, and 24-weeks post-enrollment
  Interventions: Other: STRIDE
- Medication Monitoring Control (Active Comparator): * Medication monitoring plus standard care
  * Participants will store hormonal therapy medication in a bottle provided by the study team.
  * Participants will complete questionnaires at enrollment, 12-weeks and 24-weeks post-enrollment
  Interventions: Other: Medication Monitoring Control

INTERVENTIONS:
Other: STRIDE — STRIDE is a brief, group-based, virtual (videoconference) cognitive-behavioral intervention. The intervention incorporates adherence problem-solving, cognitive restructuring, relaxation training, symptom management, coping skills training, and mindfulness techniques.
  Arms: STRIDE; STRIDE Run-In
Other: Medication Monitoring Control — Care provided as standard by the hospital and medication monitoring
  Arms: Medication Monitoring Control

SUMMARY:
The purpose of this study is to explore the feasibility and acceptability of a brief, virtual, group-based cognitive-behavioral intervention for breast cancer survivors taking hormonal therapy. The intervention (STRIDE) aims to alleviate symptoms related to hormonal therapy or breast cancer, optimize medication-taking (i.e., adherence), and reduce distress.

DETAILED DESCRIPTION:
Background: The majority of breast cancer is hormone sensitive and treated with 10 years of adjuvant endocrine therapy (AET) (i.e., tamoxifen, aromatase inhibitors) to reduce risk of recurrence and improve survival; however, adherence to AET among breast cancer survivors (BCS) is a challenge, with half of women becoming non-adherent within five years. Difficulty coping with symptoms (e.g., sleep problems, hot flashes, weight gain, fatigue) and psychosocial distress (i.e., depression or anxiety symptoms), and other emotional and logistical factors are major barriers to adherence. There is a dearth of efficacious interventions targeting the needs and adherence challenges of BCS prescribed AET.

Objective: To address this gap, the proposed study, funded by the National Cancer Institute, employs a mixed-methods design to develop and test an evidence-based intervention (STRIDE) to enhance adherence to AET, improve symptom management, and reduce distress in breast cancer survivors.

Specific Aims: The primary aims of this study are: 1) to examine the feasibility and acceptability of a tailored, small-group, virtual intervention (STRIDE) compared to a medication monitoring control for survivors of breast cancer taking AET, and 2) to explore the effects of the STRIDE intervention on adherence to AET, symptom distress, and satisfaction with AET.

Study Design: Phase 1 included (1) semi-structured interviews with BCS on AET (n=30) and intervention development with psychologists and oncology clinicians. The intervention is a a brief, virtual, small-group, cognitive-behavioral intervention that aims to alleviate symptoms and side effects related to hormonal therapy or breast cancer, optimize medication-taking, and reduce emotional distress for breast cancer survivors taking hormonal therapy. Phase 2 will entail a run-in phase (n=5) to evaluate acceptability and further refine the intervention, followed by a randomized controlled pilot trial (n=100) to assess the feasibility of comparing the STRIDE intervention to a medication monitoring control with assessments and adherence monitoring over the course of six months. Participants will be recruited at Massachusetts General Hospital Cancer Center and three community satellite sites. Eligible participants will be hormone-receptor positive breast cancer survivors prescribed AET who are experiencing distress related to AET (e.g., adherence difficulties, side effects, etc.). This research study involves completing 3 questionnaire batteries at the time of enrollment, 12 weeks, and 24 weeks. The participant will also be asked to store their hormonal therapy pills in a medication bottle provided by the study team throughout the 24 week study period. If the participants are randomized to receive the STRIDE intervention, the participant will have six weekly one-hour virtual (videoconferencing) sessions in small groups with a trained clinician followed by two 15-minute check-in phone calls later in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21 or older
* Diagnosis of early-stage (Stage 0-IIIb), hormone receptor + breast cancer
* Within 1 week-36 months of starting adjuvant endocrine therapy
* Ability to read and respond in English
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Currently taking adjuvant endocrine therapy (i.e. if took recent break, has taken within the past 2 weeks)
* Completed primary treatment (i.e., chemotherapy, surgery, and/or radiation) for early-stage breast cancer
* Indicates a score ≥4 on one of the three NCCN adapted distress thermometer study screening questions

Exclusion Criteria:

* Uncontrolled psychosis, active suicidal ideation, or psychiatric hospitalization within the past year
* Cognitive impairment that prohibits participation in the study
* Enrollment in a different clinical trial for breast cancer
* Current participation in formal group psychotherapy or other psychosocial intervention trial
* Undergoing primary treatment for other cancer (i.e., advanced stage cancer)

Min Age: 21 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M. Jacobs, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Walsh LE, Dunderdale L, Horick N, Temel JS, Greer JA, Jacobs JM. Intervention-Related Changes in Coping Ability Drives Improvements in Mood and Quality of Life for Patients Taking Adjuvant Endocrine Therapy. Psychooncology. 2024 Dec;33(12):e70049. doi: 10.1002/pon.70049. PMID 39706803
- [Derived] Walsh EA, Post K, Massad K, Horick N, Antoni MH, Penedo FJ, Safren SA, Partridge AH, Peppercorn J, Park ER, Temel JS, Greer JA, Jacobs JM. Identification of patient subgroups who benefit from a behavioral intervention to improve adjuvant endocrine therapy adherence: a randomized-controlled trial. Breast Cancer Res Treat. 2024 Apr;204(3):547-559. doi: 10.1007/s10549-023-07228-z. Epub 2024 Jan 17. PMID 38231313
- [Derived] Jacobs JM, Rapoport CS, Horenstein A, Clay M, Walsh EA, Peppercorn J, Temel JS, Greer JA. Study protocol for a randomised controlled feasibility trial of a virtual intervention (STRIDE) for symptom management, distress and adherence to adjuvant endocrine therapy after breast cancer. BMJ Open. 2021 Jan 4;11(1):e041626. doi: 10.1136/bmjopen-2020-041626. PMID 33397667

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment paused due to the COVID-19 pandemic from mid-March 2020 through May of 2020. Run-in participants were not enrolled as part of the randomized controlled trial. The purpose of the run-in arm was to trial the intervention content with participants and the purpose of any data collection in this arm was to refine the intervention content to enhance acceptability and feasibility for the RCT. Since run-in participants were not enrolled in the RCT we are not reporting these results.
Groups:
- STRIDE: * Stride is delivered as six weekly one-hour virtual (videophone) sessions in small groups with a trained clinician (or individually, in the rare instance in which scheduling doesn't allow for groups and the participant is approaching the 12-week assessment window)
  * Two 15-minute check-in phone calls later in the study
  * Participants will store hormonal therapy medication in a bottle provided by the study team.
  * Participants will complete questionnaires at enrollment, 12-weeks, and 24-weeks post-enrollment
  STRIDE: STRIDE is a brief, group-based, virtual (videoconference) cognitive-behavioral intervention. The intervention incorporates adherence problem-solving, cognitive restructuring, relaxation training, symptom management, coping skills training, and mindfulness techniques.
- Medication Monitoring Control: * Medication monitoring plus standard care
  * Participants will store hormonal therapy medication in a bottle provided by the study team.
  * Participants will complete questionnaires at enrollment, 12-weeks and 24-weeks post-enrollment
  Medication Monitoring Control: Care provided as standard by the hospital and medication monitoring
Period: Overall Study
Arm/Group | STRIDE | Medication Monitoring Control
Started | 50 | 50
Completed | 45 | 47
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STRIDE | Medication Monitoring Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 35 | 37 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.6) | 54.9 (11.2) | 56.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 47 | 47 | 94
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  African American or Black | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 47 | 44 | 91
  Other | 1 | 2 | 3
  Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Type of Adjuvant Endocrine Therapy [Count of Participants; unit: Participants]
  Aromatase Inhibitor | 28 | 32 | 60
  Tamoxifen | 22 | 18 | 40
Breast Cancer Stage [Count of Participants; unit: Participants] — Breast Cancer Stage per the AJCC Cancer Staging Manual and as determined by the treating oncologist. As the stage of breast cancer increases from zero to three, the degree of severity increases, and the patient's prognosis worsens. Stage four breast cancer indicates that breast cancer has traveled outside of the breast and regional lymph nodes to a distant organ and is considered advanced breast cancer. Patients with stage four, advanced breast cancer were not eligible for this study.
  Participants
    Stage 0 | 5 | 3 | 8
    Stage I | 36 | 41 | 77
    Stage II | 6 | 10 | 16
    Stage III | 3 | 2 | 5
Ovarian Suppression [Count of Participants; unit: Participants] — Ovarian suppression is the medical suppression of ovarian function often utilized in pre-menopausal patients with estrogen-receptor-positive breast cancer in combination with other anti-cancer therapies to lower estrogen levels. In this study, study staff determined if patients underwent ovarian suppression via chart review of the electronic medical record.
  Participants
    Receiving Ovarian Suppression | 8 | 20 | 28
    Not Receiving Ovarian Suppression | 42 | 30 | 72

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Acceptability
Description: The investigators will evaluate program feasibility by examining rates of recruitment (enrollment rate > 50%), retention (follow-up assessment completion rate > 70% of all participants who complete baseline) and attendance of program sessions (attendance rate of at least 70% of participants completing at least 4 of 6 sessions [67%]).
  The investigators will evaluate program acceptability by examining satisfaction scores on the Client Satisfaction Questionnaire (CSQ). The program will be deemed acceptable if >75% of participants report average satisfaction scores greater than the CSQ's mid-point. The CSQ is scored on a four-point Likert scale with higher scores indicating higher satisfaction.
Time Frame: 12 weeks
Population: The analysis populations are as follows.
  Feasibility:
  Enrollment - 141 eligible participants were approached and 100 participants enrolled (70.9%).
  For the remainder of the feasibility analyses, the analysis population will utilize a denominator of 100 participants enrolled to the STRIDE study.
  For the acceptability analysis, the analysis population will utilize a denominator of the 43 participants who completed at least four out of the six STRIDE sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | STRIDE | Medication Monitoring Control
Number analyzed (Participants) | 50 | 50
Participants
  Feasibility - Retention at Week 12 | 46 | 47
  Feasibility - Session Attendance | 45 | 47
  Acceptability: number analyzed (Participants) | 43 | 47
  Acceptability | 41 | NA — The Medication Monitoring Control Group did not attend intervention sessions and so did not rate acceptability.

2. Secondary Outcome: Group Differences in Mean Medication Adherence Rates to Adjuvant Endocrine Therapy Across the 24-week Study Period
Description: Medication Event Monitoring System (MEMS Caps): Participants will store medication in the MEMS bottles to electronically monitor adjuvant endocrine therapy daily dose and timing of dose administration. Prescribed medication, dose, and timing will be identified in the Electronic Health Record and verified by the patient. Adherence will be calculated as the percentage of medication taken of the total prescribed. A mean medication adherence rate will be calculated in each group to examine differences in adherence rates and changes across the 24-week study period between groups.
Time Frame: Mean medication adherence rates over 24 weeks
Population: Analysis Population includes the participants in both arms using the MEMs caps throughout the study period.
Measure: Mean (95% Confidence Interval); unit: percentage of medication taken
Arm/Group | STRIDE | Medication Monitoring Control
Number analyzed (Participants) | 45 | 47
percentage of medication taken | 84.75 [78.80 to 90.70] | 82.00 [75.98 to 88.03]
Statistical Analysis 1: Comparison: STRIDE vs Medication Monitoring Control; Analysis comparing the change in monthly adherence to adjuvant endocrine therapy across the study period adjusting for distress and receipt of ovarian suppression; Test type: Superiority; p = .504, ANCOVA — a priori threshold p<0.05; Adjusted for distress and receipt of ovarian suppression; Slope = -0.66, 95% CI 2-sided [-2.59 to 1.27]
Statistical Analysis 2: Comparison: STRIDE vs Medication Monitoring Control; Analysis comparing the change in weekly adherence rates to adjuvant endocrine therapy across the study period adjusting for distress and receipt of ovarian suppression; Test type: Superiority; p = .225, ANCOVA — a priori threshold p<0.05; Adjusted for distress and receipt of ovarian suppression; Slope = -0.17, 95% CI 2-sided [-0.44 to -0.10]

3. Secondary Outcome: Changes in Self-Reported Adjuvant Endocrine Therapy Adherence Between Groups on the Medication Adherence Report Scale (MARS-5) From Baseline to 12-weeks Post-baseline
Description: Medication Adherence Report Scale (MARS-5): Changes in self-reported adherence to adjuvant endocrine therapy between groups will be explored using the MARS-5 at 3-months post-baseline. The MARS-5 assesses adherence to treatment and has been used specifically in the context of AET adherence. The scale consists of five items that ask about suboptimal adherence behaviors, such as "I stop taking my adjuvant endocrine therapy medicine for a while." Each item is answered on a scale of 1 (Always) to 5 (Never). Scores range from 5 to 25 points with scores less than 25 defined as low adherence to the medication.
Time Frame: Baseline, and post-intervention at 12-weeks post-baseline
Population: Analysis Population includes the participants in both arms that completed the MARS-5 measure at 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | STRIDE | Medication Monitoring Control
Number analyzed (Participants) | 45 | 47
units on a scale | 23.99 [23.61 to 24.36] | 23.86 [23.49 to 24.23]
Statistical Analysis 1: Comparison: STRIDE vs Medication Monitoring Control; Analysis comparing the change in self-reported endocrine therapy adherence between groups on the MARS-5 scale from baseline to 12-weeks post-baseline adjusting for distress, receipt of ovarian suppression, and baseline values of criterion outcome; Test type: Superiority; p = .630, ANCOVA — a priori threshold p < 0.05; Adjusted for baseline values of criterion outcomes, distress and receipt of ovarian suppression; Mean Difference (Final Values) = .13, 95% CI 2-sided [-0.40 to 0.66]

4. Secondary Outcome: Changes in Satisfaction With Adjuvant Endocrine Therapy (AET) Between Groups on the Cancer Therapy Satisfaction Questionnaire (CTSQ) From Baseline to 12-weeks Post-baseline.
Description: Cancer Therapy Satisfaction Questionnaire (CTSQ): Changes in self-reported satisfaction with AET will be explored between groups at 12 weeks post-baseline with the Cancer Therapy Satisfaction Questionnaire (CTSQ). The CTSQ is a previously published 21-item measure that evaluates patients' beliefs about the following aspects of medical care: expectations of the effectiveness of cancer therapy, feelings about side effects, oral cancer therapy adherence, satisfaction with cancer therapy, stopping cancer therapy, and reasons for non-adherence. We used the satisfaction with cancer therapy subscale. Each item is scored on a scale of 1 ("Never" or "Very inconvenient") to 5 ("Always" or Very Convenient"). A greater score on this measure indicates greater patient cancer therapy satisfaction. Scores can range from a minimum of 0 to a maximum of 100.
Time Frame: Baseline, and post-intervention at 12-weeks post-baseline
Population: The analysis population includes the 92 participants in the STRIDE study who completed the CTSQ at 12 weeks.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | STRIDE | Medication Monitoring Control
Number analyzed (Participants) | 45 | 47
units on a scale | 66.53 [63.82 to 69.23] | 63.94 [61.30 to 66.58]
Statistical Analysis 1: Comparison: STRIDE vs Medication Monitoring Control; Analysis comparing the change in satisfaction with adjuvant endocrine therapy between groups on the CTSQ from baseline to 12 weeks post-baseline adjusting for distress, receipt of ovarian suppression, and baseline values of criterion outcome; Test type: Superiority; p = .186, ANCOVA — a priori threshold p < 0.05; Adjusted for baseline values of criterion outcomes, distress and receipt of ovarian suppression; Mean Difference (Final Values) = 2.58, 95% CI 2-sided [-1.27 to 6.44]

5. Secondary Outcome: Changes in Symptom Distress Between Groups on the Breast Cancer Prevention Trial Symptom Scale (BCPT) From Baseline to 12-weeks Post-baseline
Description: Breast Cancer Prevention Trial Symptom Scale (BCPT): The investigators will examine changes in self-reported symptom distress on the BCPT between groups at 12 weeks post-baseline. The BCPT is a symptom checklist used to document physical and psychological symptoms associated with ET use. The measure includes several clinically-relevant symptom subscales and has been used broadly in previous studies on symptom distress in breast cancer patients. The BCPT asks participants to rate how much they have been bothered by several symptoms over the past week on a scale of 0 (Not at all bothered) to 4 (Extremely bothered). There are 8 subscales: hot flashes, nausea, bladder control, vaginal problems, musculoskeletal pain, cognitive problems, weight problems, and arm problems. For this study, we summed the 8 subscale scores for a total score ranging from 0-72, with higher scores representing greater symptom distress.
Time Frame: Baseline and post-intervention at 12 weeks post-baseline
Population: The analysis population includes the 92 participants in the STRIDE study who completed the BCPT at 12 weeks.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | STRIDE | Medication Monitoring Control
Number analyzed (Participants) | 45 | 47
units on a scale | 19.89 [17.98 to 21.79] | 20.67 [18.82 to 22.53]
Statistical Analysis 1: Comparison: STRIDE vs Medication Monitoring Control; Analysis comparing the change in symptom distress between groups on the BCPT scale from baseline to 12-weeks post-baseline adjusting for distress, receipt of ovarian suppression, and baseline values of criterion outcome; Test type: Superiority; p = .562, ANCOVA — a priori threshold p < 0.05; Adjusted for baseline values of criterion outcomes, distress and receipt of ovarian suppression; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-3.49 to 1.91]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | STRIDE | Medication Monitoring Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Study recruitment paused due to the COVID-19 pandemic from mid-March 2020 through May of 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT03837496/Prot_SAP_000.pdf